CLINICAL TRIAL: NCT03302156
Title: PSMA Positron Emission Tomography (PET) and Magnetic Resonance (MR) Imaging in Gynecological Cancers
Brief Title: PSMA PET and MRI in Gynecological Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual following suspension per COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UW17017; 2017-0456 (Other: Institutional Review Board); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison); NCI-2018-00466 (Registry Identifier: NCI Trial ID); 06-08-2020 (Other: Protocol Version Date)
Record Dates: First submitted 2017-08-18; First posted 2017-10-04 (Actual); Results first posted 2023-08-09 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-07

CONDITIONS: Gynecologic Cancer
Keywords: Uterine cancer; Ovarian cancer; Hysterectomy; Salpingo-oophorectomy
MeSH Terms: conditions — Uterine Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Control Non-Dosimetry Group (Other): The control group will consists of women with no imaging evidence of gynecological cancer, who are undergoing hysterectomy and salpingo-oophorectomy. Women will receive PSMA-based 18F-DCFPyL tracer and PET/MR imaging. n=6
  Interventions: Drug: PSMA-based 18F-DCFPyL PET tracer
- Patient Group (Other): The patient group will consist of women with suspected gynecological cancers who are undergoing hysterectomy and salpingo-oophorectomy. Women will receive standard of care PSMA-based 18F-DCFPyL tracer and PET/MR imaging. n=40
  Interventions: Drug: PSMA-based 18F-DCFPyL PET tracer
- Dosimetry Group (Other): Women with or without suspected gynecological cancer. Women will receive PSMA-based 18F-DCFPyL tracer and PET/CT imaging, PET/MR imaging as needed. n=6
  Interventions: Drug: PSMA-based 18F-DCFPyL PET tracer

INTERVENTIONS:
Drug: PSMA-based 18F-DCFPyL PET tracer — PSMA-based 18F-DCFPyL PET tracer that will be used to determine the presence or absence of cancer
  Other Names: PSMA

SUMMARY:
The goal of this research is to determine the accuracy of PSMA positron emission tomography (PET) and multi-parametric magnetic resonance (MR) imaging to detect the presence of gynecological cancer cells in the body.

DETAILED DESCRIPTION:
The investigators will evaluate a novel second-generation low-molecular-weight prostate specific membrane antigen (PSMA)-based positron emission tomography (PET) agent, 18F-DCFPyL, to determine the presence or absence of cancer, the accurate distribution of cancer and the normal biodistribution of PSMA in the abdomen and pelvis on PET imaging.

PSMA, also known as folate hydrolase 1 and glutamate carboxypeptidase II, is an enzyme associated with prostate cancer but has been also found to be expressed in the tumor neovasculature of many different types of non-prostate cancer tumors. PSMA-based 18F-DCFPyL PET demonstrates very high tumor-to-background ratio when studied in other tumors, including prostate tumors.

MR imaging is a highly sensitive and specific imaging modality that can be used for gynecologic cancers. MR images can be obtained in conjunction with PSMA PET, adding additional anatomic and multi-parametric MRI information without the need for a second imaging appointment.

ELIGIBILITY:
Inclusion Criteria for healthy female controls N=12 (includes up to 6 Dosimetry participants):

* Women with no suspected gynecological cancer.
* No contraindications for MR or PET imaging.
* Greater than or equal to 18 years of age.
* Scheduled to undergo a hysterectomy and/or salpingo-oophorectomy

Inclusion Criteria for female controls (Dosimetry):

* Women with or without suspected gynecological cancer.
* No contraindications for MR or PET imaging.
* Greater than or equal to 18 years of age.

Inclusion Criteria for gynecological cancer patients (N=40):

* Women with known or suspected gynecological cancer
* No contraindications for MR or PET imaging.
* Greater than or equal to 18 years
* Have had or are scheduled to undergo a hysterectomy and/or salpingo-oophorectomy

Exclusion Criteria:

* Women that are pregnant or breast-feeding.
* Age <18
* Inability to provide informed consent on their own behalf
* Severe kidney dysfunction (GFR <30 mL/min/1.73m2)

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Cho, MD, Principal Investigator — University of Wisconsin, Madison; Elizabeth Sadowski, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Kunikowska J, Bizon M, Pelka K, Derlatka P, Olszewski M, Krolicki L. 68 Ga-Prostate-Specific Membrane Antigen PET/CT in Ovarian Tumors : Potential to Differentiate Benign and Malignant Tumors Before Surgery: A Preliminary Report. Clin Nucl Med. 2023 Feb 1;48(2):e60-e66. doi: 10.1097/RLU.0000000000004486. Epub 2022 Nov 18. PMID 36512649
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 15 participants were consented from November 2017 to December 2019. Research was suspended in March 2020 per the COVID-19 pandemic. The study opened to enrollment again in June 2022; there were no more participants consented. The investigator terminated the study in January 2023 due to slow accrual of patients with ovarian cancer and due to lack of funding. No participants were enrolled in the Dosimetry group.
Period: Overall Study
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Dosimetry Group
Started | 2 | 13 | 0
Analysis Population | 2 | 12 | 0
Participants With Confirmed Ovarian Cancer With PSMA Uptake | 0 | 1 | 0
Completed | 2 | 12 | 0
Not Completed | 0 | 1 | 0
Not completed — no visible evidence of tumor on MRI | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: study terminated early, no participants enrolled in dosimetry group
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Total
Number analyzed (Participants) | 2 | 12 | 14
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [39 to 68] | 57.3 [36 to 86] | 56.7 [36 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 12 | 14
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 12 | 14
Suspected Participant Diagnosis [Count of Participants; unit: Participants]
  Healthy Controls | 2 | 0 | 2
  Ovarian Cancer | 0 | 8 | 8
  Endometrial Cancer | 0 | 3 | 3
  Cervical Cancer | 0 | 0 | 0
  Other Cancer | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Accuracy
Description: Estimate the frequency with which PSMA PET and MR imaging and final IHC staining disagree in their classifications of presence of disease.
Time Frame: up to 1 day
Population: Calculating accuracy relies on the IHC staining as the gold standard. IHC staining was not done because the study was terminated due to low recruitment and loss of funds. Because the IHC staining was not performed, there is no gold standard by which to perform accuracy, sensitivity and specificity analysis.
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Dosimetry Group
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Biodistribution of PSMA Measured by SUVmax in Normal Tissue
Description: Record the normal biodistribution of PSMA as detected in normal tissue controls, by the resulting PET imaging.
Time Frame: up to 1 day
Population: This was performed on the entire population of patients recruited in both the Healthy Control and Patient group.
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Dosimetry Group
Number analyzed (Participants) | 2 | 12 | 0
SUVmax
  Aorta at carina | 2.0 (0.1) | 1.7 (0.5) |
  Liver - Right Lobe | 12.1 (5.4) | 10.0 (0.5) |
  Myometrium: number analyzed (Participants) | 2 | 9 | 0
  Myometrium | 2.2 (0.4) | 2.9 (0.5) |
  Endometrium: number analyzed (Participants) | 2 | 7 | 0
  Endometrium | 5.9 (1.8) | 4.8 (0.5) |
  Cervix: number analyzed (Participants) | 2 | 8 | 0
  Cervix | 4.0 (1.1) | 3.3 (0.5) |
  Right Ovary: number analyzed (Participants) | 2 | 5 | 0
  Right Ovary | 1.5 (1.7) | 3.0 (0.5) |
  Corpus Luteum: number analyzed (Participants) | 1 | 3 | 0
  Corpus Luteum | 6.3 (NA) — Standard deviation was not calculated as only a single participant was analyzed | 5.9 (0.5) |
  Left Ovary: number analyzed (Participants) | 2 | 5 | 0
  Left Ovary | 1.7 (1.4) | 2.3 (0.5) |

3. Secondary Outcome: Biodistribution of PSMA Measured by SUVmax in Cancer Tissue
Description: Record the biodistribution of PSMA as detected in cancer tissue, by the resulting PET imaging.
Time Frame: up to 1 day
Population: This was performed on the "Patient" population. There was only one patient with confirmed ovarian cancer with PSMA uptake.
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Dosimetry Group
Number analyzed (Participants) | 0 | 1 | 0
SUVmax |  | 10.5 (NA) — Standard deviation was not calculated as only a single participant was analyzed |

4. Secondary Outcome: Radiodosimetry of PSMA
Description: The radiodosimetry of PSMA-based 18F-DCFPyL will be measured in normal female controls via the resulting PET images.
Time Frame: up to 1 day
Population: No data was collected for this. There were no participants enrolled into the Dosimetry group. The study was terminated early due to low accrual and loss of funding.
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Dosimetry Group
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Sensitivity and Specificity of PSMA-based PET/MR
Description: Record the distribution of PSMA in cancer tissue.
Time Frame: up to 1 day
Population: Calculating sensitivity and specificity relies on the IHC staining as the gold standard. IHC staining was not done because the study was terminated due to low recruitment and loss of funds. Because the IHC staining was not performed, there is no gold standard by which to perform accuracy, sensitivity and specificity analysis.
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group | Dosimetry Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: during research visit, up to 3 hours
Arm/Group | Healthy Control Non-Dosimetry Group | Patient Group
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/12
Other Adverse Events (participants affected / at risk) | 0/2 | 0/12

LIMITATIONS AND CAVEATS:
Calculating accuracy, sensitivity and specificity relies on the IHC staining as the gold standard. IHC staining was not done because the study was terminated due to low recruitment and loss of funds. Because the IHC staining was not performed, there is no gold standard by which to perform accuracy, sensitivity and specificity analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT03302156/Prot_SAP_000.pdf